CLINICAL TRIAL: NCT05065502
Title: Maintaining Implementation Through Dynamic Adaptations (MIDAS) (QUE 20-025)
Brief Title: MIDAS Cluster Randomized Controlled Trial of Implementation Strategies to Optimize Use of Medications in VA Clinical Settings
Acronym: MIDAS cRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: QUX 21-004
Record Dates: First submitted 2021-08-17; First posted 2021-10-04 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Polypharmacy; Insomnia; Anticoagulants
Keywords: implementation science; implementation strategy; anticoagulation; polypharmacy; insomnia; medication safety; academic detailing; quality improvement; pragmatic trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The investigators will conduct a series of three trials to test two implementation strategies designed for sustained change. Each trial will be a two-arm, cluster-randomized trial. The results of these trials will be pooled together in a single cross-trial analysis using a dichotomous outcome for each trial. Each trial will also be analyzed independently. Two of the trials will use the same dichotomous primary outcome and the third trial will use a different primary outcome (CBTI). The two arms will both include use of clinical population health dashboards. Unit of analysis is clinic. Clinics will be randomized to one of two implementation strategies described below. Implementation strategies will be tested for effectiveness of sustained use of practices to address documented quality gaps related to (1) potentially inappropriate medications, (2) use of direct oral anticoagulation medications (DOACs), and (3) cognitive behavioral therapy as first-line treatment for insomnia (CBTI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Academic Detailing (AD) Only (Active Comparator): One-on-one educational outreach to employees and providers.
  Interventions: Behavioral: Academic Detailing (AD)
- AD + LEAP Combined (Experimental): This arm combines use of AD plus the Learn. Engage. Act. Process (LEAP) program. LEAP is a 6-month quality improvement coaching program plus a 6-month monthly follow-up.
  Interventions: Behavioral: Academic Detailing (AD); Behavioral: LEAP

INTERVENTIONS:
Behavioral: Academic Detailing (AD) — The National Resource Center for Academic Detailing (NaRCAD) describes AD as "an innovative, one-on-one outreach education technique that helps clinicians provide evidence-based care to their patients. Using an accurate, up-to-date synthesis of the best clinical evidence in an engaging format, academic detailers ignite clinician behavior change, ultimately improving patient health. A successful AD visit is highly interactive, always a dialogue, and assesses a clinician's individual needs, beliefs, attitudes, issues, and concerns in order to promote better.[practice]."
Behavioral: LEAP — Learn. Engage. Act. Process (LEAP) program is a structured 6-month core curriculum plus 6 monthly collaborative sessions. The LEAP quality improvement program engages frontline teams in sustained incremental improvements of EBPs over a six-month period, allowing space for busy clinicians to learn and immediately apply fundamental QI skills. LEAP encompasses: 1) a structured, accessible curriculum based on the Institute for Healthcare Improvement's (IHI) Model for Improvement and Plan-Do-Study-Act cycles of change; 2) team-based, hands-on learning, and 3) coaching support and a QI network to enhance learning and accountability.
  Arms: AD + LEAP Combined

SUMMARY:
Scientific advances are constantly leading to better treatments. However, it is quite challenging for healthcare systems, including VA, to ask very busy providers to change the way they practice. The MIDAS QUERI program will help providers improve the way they treat VA patients for three common conditions, using specific strategies to ensure the reliable delivery of these treatments. The first project will focus on reducing potentially inappropriate medication (PIM) use using the VIONE practice, developed in VA. The second project will focus on better use of drugs called direct oral anticoagulants (DOACs) for patients with a history of severe blood clots or an abnormal heart rhythm. The third project will focus on increasing the use of cognitive behavioral therapy for insomnia as the first-line treatment for insomnia instead of sleep medications. The investigators will test two implementation approaches to improve medication use within these topics.

DETAILED DESCRIPTION:
Background The adoption and sustainment of evidence-based practices (EBPs) is a challenge within many healthcare systems, especially in settings that have already strived but failed to achieve longer-term goals. The Veterans Affairs (VA) Maintaining Implementation through Dynamic Adaptations (MIDAS) Quality Enhancement Research Initiative (QUERI) program was funded as a series of trials to test multi-component implementation strategies to sustain optimal use of three EBPs: 1) a deprescribing approach intended to reduce potentially inappropriate polypharmacy; 2) appropriate dosing and drug selection of direct-acting anticoagulant medications (DOACs); and 3) use of cognitive behavioral therapy as first-line treatment for insomnia before pharmacologic treatment. We describe the design and methods for a harmonized series of cluster-randomized control trials comparing two implementation strategies.

Methods For each trial, we will recruit 8-12 clinics (24-36 total). All will have access to a clinical dashboard that flags patients who may benefit from the target EBP at that clinic and provider. For each trial, clinics will be randomized to one of two implementation strategies to improve use of the EBPs: 1) individual-level academic detailing (AD); or 2) AD plus the team-based Learn. Engage. Act. Process. (LEAP) quality improvement (QI) learning program. The primary outcomes will be operationalized across the three trials as a patient-level dichotomous response (yes/no) indicating patients with potentially inappropriate medications (PIMs) among those who may benefit from the EBP. This outcome will be computed using month-by-month administrative data. Primary comparison between the two implementation strategies will be analyzed using generalized estimating equations (GEE) with clinic-level monthly percent of PIMs as the dependent variable. Primary comparative endpoint will be at 13-18 months post-baseline. Each trial will also be analyzed independently.

Discussion MIDAS QUERI trials will focus on fostering sustained use of EBPs that previously had targeted but incomplete implementation. Our implementation approaches are designed to engage frontline clinicians in a dynamic optimization process that integrates use of actionable clinical dashboard data and making incremental changes, designed to be feasible within busy clinical settings.

ELIGIBILITY:
Inclusion Criteria:

Note- the investigators are recruiting clinics - not individual patients.

* Prior to implementation, the investigators will work with sites to ensure they have met the preconditions necessary to begin sustained optimization of the EBP:

  * a team leader or champion
  * an identified department with service leadership buy-in and control over the processes/practices impacted by the implementation
  * readily accessible data to measure process and impact of the implementation and use of the EBP
  * availability of required resources

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy B. Sussman, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Ariel Domlyn, PhD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Jacob E Kurlander, MD MS MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Paul N Pfeiffer, MD MS, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Site-level data that underlie results reported, after de-identification will be available.
Supporting Information: Study Protocol, Analytic Code
Time Frame: For 36 months after article is published.
Access Criteria: Upon request by researchers who provide a methodologically sound proposal. Further details will be available.

REFERENCES:
- [Derived] Domlyn AM, Hooks G, Freitag M, Evans L, Stewart M, Damschroder L, Sussman JB. Core and modifiable components of academic detailing: demonstration of implementation strategy development, tailoring, and documentation process. Front Health Serv. 2025 Jun 3;5:1521504. doi: 10.3389/frhs.2025.1521504. eCollection 2025. PMID 40529793
- [Derived] Damschroder LJ, Sussman JB, Pfeiffer PN, Kurlander JE, Freitag MB, Robinson CH, Spoutz P, Christopher MLD, Battar S, Dickerson K, Sedgwick C, Wallace-Lacey AG, Barnes GD, Linsky AM, Ulmer CS, Lowery JC. Maintaining Implementation through Dynamic Adaptations (MIDAS): protocol for a cluster-randomized trial of implementation strategies to optimize and sustain use of evidence-based practices in Veteran Health Administration (VHA) patients. Implement Sci Commun. 2022 May 14;3(1):53. doi: 10.1186/s43058-022-00297-z. PMID 35568903

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: VA medical centers and/or clinics
Groups:
- Academic Detailing (AD) Only: Academic Detailing (AD): Site providers received one-on-one educational sessions between a non-physician professional trained in communication skills and the specific topic area (the Academic Detailer) aimed at increasing the use of the evidence-based practices.
- AD + LEAP Combined: Academic Detailing (AD): Site providers received one-on-one educational sessions between a non-physician professional trained in communication skills and the specific topic area (the Academic Detailer) aimed at increasing the use of the evidence-based practices.
  LEAP: Sites also received the Learn. Engage. Act. Process. (LEAP) program, which is a 6-month quality improvement coaching program plus a 6-month follow-up.
Period: Overall Study
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Started | NA; 14 VA medical centers and/or clinics (The intervention was completed at the facility level.) | NA; 14 VA medical centers and/or clinics (The intervention was completed at the facility level.)
Completed | NA; 12 VA medical centers and/or clinics (The intervention was completed at the facility level.) | NA; 12 VA medical centers and/or clinics (The intervention was completed at the facility level.)
Not Completed | NA; 2 VA medical centers and/or clinics | NA; 2 VA medical centers and/or clinics

BASELINE CHARACTERISTICS:
Population: These numbers refer to all individuals who were eligible for each EBP at the baseline of the clinical trial.
Units Other Than Participants: VA medical centers and/or clinics
Groups:
- Total: Total of all reporting groups
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined | Total
Number analyzed (Participants) | 79481 | 66208 | 145689
Number analyzed (VA medical centers and/or clinics) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The row population differs from the overall population because age was missing for some participants
  years
    number analyzed (Participants) | 79471 | 66204 | 145675
    (all) | 66.7 (16.4) | 66.3 (15.9) | 66.5 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The row population differs from the overall population because sex was missing for some participants
  Participants
    number analyzed (Participants) | 79471 | 66204 | 145675
    Female | 5201 | 4162 | 9363
    Male | 74270 | 62042 | 136312
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17593 | 2078 | 19671
  Not Hispanic or Latino | 59993 | 62991 | 122984
  Unknown or Not Reported | 1895 | 1139 | 3034
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 61865 | 51216 | 113081
  Black | 9278 | 6142 | 15420
  Asian | 546 | 1552 | 2098
  Hawaiian-Pacific | 527 | 563 | 1090
  Native-American/Alaskan Native | 432 | 746 | 1178
  Missing | 6833 | 5989 | 12822
Percent of Patients with Overall Inappropriate Medications across trials and facilities at Baseline [Mean (Standard Deviation); unit: Percent of patients with PIMs] — Percentage of Patients with Potentially Inappropriate Medication use (PIMs) across all three trials/evidence based practices (EBPs) and Facilities, at baseline.
  Percent of patients with PIMs | 12.7 (17.1) | 14.1 (19.1) | 13.4 (16.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in the Percentage of Patients With Potentially Inappropriate Medication Use (PIMs) Between Pre- and Post-periods, Across Facilities.
Description: Percentage of PIMs across AD vs. LEAP+AD facilities were modelled as the difference between post-period and pre-period, using the average from the 1-6-month pre-baseline period as "pre" and the average 13-18-month post-baseline as "post." Data was collected monthly at patient level and collapsed by clinic-month for patients who are at risk of potentially inappropriate medication use. Clinic-month outcome was computed as: 1) VIONE; proportion of patients who possessed one or more medications from the Beers' list of patients 65 or older, actively following with the clinic, and not in hospice/palliative care; 2) DOACs; proportion of patients with flags for potentially inappropriate use on a DOAC safety dashboard of those using DOACs; 3) CBTI; proportion of patients with a new prescription for a sleep medication for insomnia who have not had CBTI of those who are actively followed by the clinic and not in hospice/palliative care. The outcome was analyzed by pooling across all three-EBPs.
Time Frame: 13-18 months post-baseline
Population: The number of participants analyzed refers to all individuals who were eligible for the cross sectional analysis at any time point in the study .
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients with PIMs
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 120,891 | 96,117
Number analyzed (VA medical centers and/or clinics) | 12 | 12
percentage of patients with PIMs | -0.133 [-0.481 to 0.2144] | -0.395 [-0.800 to 0.0104]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in proportion of PIMs of post-intervention period (months 13 to 18), controlling for use in pre-baseline period (months 0 to 6), averaged across three studies; Test type: Superiority; p = 0.273, Regression, Linear — Significance level is set at 0.05; Mean Difference (Net) = -0.261, 95% CI 2-sided [-0.728 to 0.206], Standard Error of Mean 0.238 — Between-arm difference at 13-18 months post-baseline, controlling for rates 1-6 months pre-baseline

2. Secondary Outcome: Change in Patients With Percentage of Potentially Inappropriate Use of Medications (PIMs) Across Facilities
Description: Medications include proton pump inhibitors (PPIs), aspirin, central nervous system (CNS) active medications (muscle relaxants, anti-psychotics, Z-drugs, and benzodiazepines), or anticholinergic drugs. This is the primary outcome for the VIONE trial when analyzed as a stand-alone trial and the VIONE sub-analysis of the overall MIDAS study primary outcome. Percentage of patients with PIMs across AD vs. LEAP+AD facilities were modelled longitudinally using Generalized Estimating Equations (GEE), with a three way-interaction of arm, month of follow-up, and pre-, post-period. Data will was be collected monthly at patient level and collapsed by clinic-month for patients who are at risk of potentially inappropriate medication use. Estimates computed using least squares (LS) means from the GEE model.
Time Frame: 13-18 months post-baseline
Population: The number of participants refers to all individuals who were eligible for the cross sectional analysis at any time point in the VIONE study.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients with PIMs
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 19,369 | 8,130
Number analyzed (VA medical centers and/or clinics) | 6 | 6
percentage of patients with PIMs | -0.01756 [-0.03052 to -0.00459] | -0.01618 [-0.03854 to 0.00619]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in proportion of PIMs for the post-intervention period (months 13 to 18), controlling for the pre-baseline period (months 0 to 6); Test type: Superiority; Mean Difference (Net) = 0.00138, 95% CI 2-sided [-0.0245 to 0.0272]

3. Secondary Outcome: Change in Monthly Medication Costs for All Drugs Across Facilities
Description: Cost of all drugs without regard to appropriateness. Average monthly cost per patient across LEAP vs. LEAP + AD facilities were modelled longitudinally with a Generalized Linear Model with a Gamma Link and a three-way interaction of arm, month of follow-up and pre-, post-period. Estimates computed using LS means from the GEE model. This will be a secondary outcome for the VIONE trial when analyzed as a stand-alone trial.
Time Frame: 13-18 months post-baseline
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: dollars per patient
Units Other Than Participants: VA medical centers and/or clinics
Groups:
- AD + LEAP Combined: Academic Detailing (AD): Site providers received one-on-one educational sessions between a non-physician professional trained in communication skills and the specific topic area (the Academic Detailer) aimed at increasing the use of the evidence-based practices.
  LEAP: Sites also received the Learn. Engage. Act. Process. (LEAP) program, which is a 6-month quality improvement coaching program plus a 6-month follow-up. =
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 19,369 | 8,130
Number analyzed (VA medical centers and/or clinics) | 6 | 6
dollars per patient | 70.73 [34.94 to 106.52] | 13.72 [-29.76 to 57.19]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in medication costs from 6-months pre-baseline period to 6-month post-intervention period (months 13 to 18); Test type: Superiority; Mean Difference (Net) = 23, 95% CI 2-sided [-23.3 to 69.3] — Statistical Assumptions for Valid Inference of a typical Difference-in-Difference model were not met, Estimate computed from modelling Post-period, and adjusting for Pre-period

4. Secondary Outcome: Change in Number of Medication Reviews Across Facilities
Description: Number of medication reviews completed by a pharmacist. This will be a secondary outcome for the VIONE trial when analyzed as a stand-alone trial.
Time Frame: 13-18 months post-baseline
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: number of medication reviews
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 19,369 | 8,130
Number analyzed (VA medical centers and/or clinics) | 6 | 6
number of medication reviews | -0.00004 [-0.00011 to 0.00002] | -0.00064 [-0.00112 to -0.00017]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in count of medication note reviews from 6-months pre-baseline period to 6-month post-intervention period (months 13 to 18); Test type: Superiority; Median Difference (Net) = -0.599, 95% CI 2-sided [-1.080 to -0.122]; Medication reviews per 1,000 patients (outcome multiplied by 1,000). Statistical Assumptions for Valid Inference of a typical Difference-in-Difference model were not met, Estimate computed from modelling Post-period, and adjusting for Pre-period

5. Secondary Outcome: Change in Number of Inappropriate Medications at a Patient-level
Description: This is a measure of count of medications used at the patient (not facility) level. This will be a secondary outcome for the VIONE trial when analyzed as a stand-alone trial.
Time Frame: 13-18 months post-baseline
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients with PIMs
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 19369 | 8130
Number analyzed (VA medical centers and/or clinics) | 6 | 6
percentage of patients with PIMs | -0.00625 [-0.03369 to 0.02118] | -0.05942 [-0.08509 to -0.03376]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in count of inappropriate use from 6-months pre-baseline period to 6-month post-intervention period (months 13 to 18); Test type: Superiority; Mean Difference (Net) = -0.05317, 95% CI 2-sided [-0.09073 to 0.01561]

6. Secondary Outcome: Change in Percentage of Patients With High-risk Direct Oral Anticoagulant (DOAC) Use Across Facilities
Description: High-risk DOAC use will be assessed by "flags" using the algorithm from an operations DOAC dashboard. These flags were developed based on existing guidelines and advice of many anticoagulation experts. Percentage of patients with PIMs across AD vs. LEAP+AD facilities were modelled longitudinally using Generalized Estimating Equations, with a three way-interaction of arm, month of follow-up, and pre-, post-period. Data will was be collected monthly at patient level and collapsed by clinic-month for patients who are at risk of potentially inappropriate medication use. Estimates computed using LS means from the GEE model. This is the primary outcome for the DOAC trial when analyzed as a stand-alone trial and the DOAC sub-analysis of the overall MIDAS study primary outcome.
Time Frame: 13-18 months post-baseline
Population: The number of participants refers to all individuals who were eligible for the cross sectional analysis at any time point in the DOAC study.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients with a DOAC flag
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 17398 | 14495
Number analyzed (VA medical centers and/or clinics) | 4 | 4
percentage of patients with a DOAC flag | 0.64 [-0.38 to 1.66] | 0.53 [-0.32 to 1.37]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in proportion of high-risk DOAC use from 6-months pre-baseline period to 6-month post-intervention period (months 13 to 18); Test type: Superiority; Mean Difference (Net) = -0.12, 95% CI 2-sided [-1.44 to 1.20]

7. Secondary Outcome: Change in Percentage of Patients With Direct Oral Anticoagulant (DOAC) Flags Attributable to Chronic Kidney Disease Across Facilities
Description: This was the subset of patients with DOAC Population Health Management Tool (Dashboard) flags that occur when medications are given at doses that would be appropriate but are not because the patient has abnormal renal function. This has had minimal adjustments since being described in previous publications.
Time Frame: 13-18 months post-baseline
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients with a DOAC flag
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 17398 | 14495
Number analyzed (VA medical centers and/or clinics) | 4 | 4
percentage of patients with a DOAC flag | 0.31 [-0.12 to 0.75] | 0.11 [-0.33 to 0.55]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in proportion of of high-risk DOAC use attributable to chronic kidney disease for the post-intervention period (months 13 to 18), controlling for the pre-baseline period (months 0 to 6), ), controlling for the pre-baseline period (months 0 to 6); Test type: Superiority; Mean Difference (Net) = -0.20, 95% CI 2-sided [-0.83 to 0.42]

8. Secondary Outcome: Change in Percentage of Patients With Direct Oral Anticoagulant (DOAC) Flags Attributable to Weight Across Facilities
Description: This was the subset of patients with DOAC Population Health Management Tool (Dashboard) flags that occur when medications are given at doses that would be appropriate but are not because the patient has unusually high or low weight or BMI. This has had minimal adjustments since being described in previous publications.
Time Frame: 13-18 months post-baseline
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients with a DOAC flag
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 17398 | 14495
Number analyzed (VA medical centers and/or clinics) | 4 | 4
percentage of patients with a DOAC flag | 0.17 [-0.13 to 0.47] | 0.49 [0.22 to 0.76]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in proportion of high-risk DOAC use attributable to weight for the post-intervention period (months 13 to 18), controlling for the pre-baseline period (months 0 to 6); Test type: Superiority; Mean Difference (Net) = 0.32, 95% CI 2-sided [-0.08 to 0.72]

9. Secondary Outcome: Change in Percentage of Patients With Direct Oral Anticoagulant (DOAC) Flags Attributable to Other Mis-dosing Across Facilities
Description: These are the remaining high-risk flags and are usually due to patients with medication interactions or doses that are incorrect due to the indication. This has had minimal adjustments since being described in previous publications.
Time Frame: 13-18 months post-baseline
Population: as for outcome 6
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients with a DOAC flag
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 17398 | 14495
Number analyzed (VA medical centers and/or clinics) | 4 | 4
percentage of patients with a DOAC flag | 0.20 [-0.18 to 0.57] | 0.02 [-0.34 to 0.37]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in proportion of high-risk DOAC use attributable to mis-dosing for the post-intervention period (months 13 to 18), controlling for the pre-baseline period (months 0 to 6); Test type: Superiority; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.70 to 0.33]

10. Secondary Outcome: Change in Percentage of Patient Receipt of Any Cognitive Behavioral Therapy for Insomnia (CBTI) Across Facilities
Description: Patient receipt of any CBTI will be measured by extracting from the medical records CBTI note templates completed by CBTI therapists. The denominator will consist of primary care patients who are not in hospice/palliative care. Percentage of PIMs across AD vs. LEAP+AD facilities were modelled longitudinally using Generalized Estimating Equations, with a three way-interaction of arm, month of follow-up, and pre-, post-period. Data will was be collected monthly at patient level and collapsed by clinic-month for patients who are at risk of potentially inappropriate medication use. Estimates computed using LS means from the GEE model. This will be the primary outcome for the CBTI trial when analyzed as a stand-alone trial.
Time Frame: 13-18 months post-baseline
Population: The number of participants refers to all individuals who were eligible for the cross sectional analysis at any time point in the CBT-I study.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients receiving CBTI
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 90,307 | 78,842
Number analyzed (VA medical centers and/or clinics) | 4 | 4
percentage of patients receiving CBTI | -0.00922 [-0.04200 to 0.02355] | 0.00085 [-0.00898 to 0.01067]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Between group comparison is done using between-arm difference (as 'AD+LEAP' minus 'AD only') in within-arm change in proportion of CBTI receipt for the post-intervention period (months 13 to 18), controlling for the pre-baseline period (months 0 to 6); Test type: Superiority; Mean Difference (Net) = 0.01007, 95% CI 2-sided [-0.02415 to 0.04429]

11. Secondary Outcome: Change in Mean Cognitive Behavioral Therapy for Insomnia (CBTI) Sessions Completed
Description: Mean number of sessions will be measured by extracting from the medical records CBTI note templates completed by CBTI therapists. The denominator will consist of primary care patients who are not in hospice/palliative care. This will be a secondary outcome for the CBTI trial when analyzed as a stand-alone trial.
Time Frame: 13-18 months post-baseline
Population: After conducting additional testing of our algorithm for detecting CBTI sessions, we found the algorithm to be adequately sensitive to detecting *any* CBTI but not accurate for detecting the number of CBTI sessions (e.g., CBTI could often be mentioned in the context of a referral or some other ongoing treatment).
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Change in the Monthly Percentage of Patients Referred to Cognitive Behavioral Therapy for Insomnia (CBTI) Across Facilities
Description: CBTI referrals will be measured according to counts of CBTI consult requests in the medical record. For clinics that do not use medical record consult requests specific to CBTI, referrals will be measured using monthly counts provided by CBTI therapists. The denominator will consist of primary care patients who are not in hospice/palliative care. This will be a secondary outcome for the CBTI trial when analyzed as a stand-alone trial.
Time Frame: 13-18 months post-baseline
Population: It was originally planned for all CBTI sites to provide information regarding where in the medical records the investigators could identify referrals. However, prior to launching the trial, it was determined several of the sites' processes for referrals were not distinguishable as referrals vs. other forms of communication (e.g., adding a therapist as a cosigner to a note), making collection of this data impractical and not conducted. Thus, we did not have any sites collect referral information.
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Change in Percentage of Patients With First Line Sleep Medication Across Facilities
Description: The proportion of patients with a new prescription for a sleep medication for insomnia who have not had CBTI of those who are actively followed by the clinic and not in hospice/palliative care. This is a CBTI sub-analysis of the overall MIDAS study primary outcome.
Time Frame: 13-18 months post-baseline
Population: The number of participants refers to all individuals who were eligible for the cross sectional analysis at any time point in the CBTI study.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of patients PIMs
Units Other Than Participants: VA medical centers and/or clinics
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 90,307 | 78,842
Number analyzed (VA medical centers and/or clinics) | 4 | 4
percentage of patients PIMs | 0.02206 [-0.06155 to 0.10567] | -0.06164 [-0.15650 to 0.03322]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; Mean Difference (Net) = -0.0837, 95% CI 2-sided [-0.21014 to 0.04275]

14. Other Pre Specified Outcome: Change in Employee Engagement in Quality Improvement
Description: 3-item pilot measure of the extent to which employees engage in quality improvement activities given both at baseline and 18-months post-implementation. Scores are 1-5 with higher ratings indicating more engagement in quality improvement.
Time Frame: 18-months Post-baseline
Population: The number of participants refers to those eligible for AD and/or LEAP participation at baseline and those who participated in AD and/or LEAP at post-implementation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 65 | 69
units on a scale | 0.305 [-0.242 to 0.852] | 0.247 [-0.306 to 0.801]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Test type: Superiority; Mean Difference (Net) = 0.102, 95% CI 2-sided [-0.216 to 0.420]

15. Other Pre Specified Outcome: Change in Employee Burnout
Description: 3-item measure comprising one item each for exhaustion, depersonalization, and reduced achievement (reverse scored) given both at baseline and 18-months post-implementation. "High Burnout" measures the percent of staff who are feeling burned out on all three burnout items at a frequency of "once a week" to "every day." Scored: 0-100%, where LOWER score is more favorable.
Time Frame: 18-months post-baseline
Population: The number of participants refers to those eligible for AD and/or LEAP participation at baseline and/or those who participated in AD and/or LEAP at post-implementation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 67 | 70
units on a scale | -0.586 [-1.298 to 0.127] | 0.227 [-0.441 to 0.895]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Test type: Superiority; Mean Difference (Net) = -0.0389, 95% CI 2-sided [-0.555 to 0.477]

16. Other Pre Specified Outcome: Change in Best Places to Work Score
Description: 3-item scale. "Best Places to Work" (BPTW) is a summary measure of the group's satisfaction with the job, organization, and likelihood to recommend VA as a good place to work given both at baseline and 18-months post-implementation. The values are 1 to 5 with a higher score being more positive and the BPTW score is the average of the 3 questions. This is a measure normally administered within the All-employee Survey (AES) and the questions come from the Partnership for Public Service's BPTW survey (http://bestplacestowork.org).
Time Frame: 18-months post-baseline
Population: as for outcome 14
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 67 | 71
units on a scale | 0.170 [-0.412 to 0.752] | -0.056 [-0.636 to 0.524]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Test type: Superiority; Mean Difference (Net) = 0.101, 95% CI 2-sided [-0.250 to 0.452]

17. Other Pre Specified Outcome: Change in Workgroup Cohesion & Engagement
Description: 7-item measure from the VA's newly developed Patient Safety Culture given both at baseline and 18-months post-implementation. Values 1 to 5 where higher values indicate more positive scores.
Time Frame: 18-months post-baseline
Population: as for outcome 15
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
Number analyzed (Participants) | 67 | 68
units on a scale | 0.131 [-0.348 to 0.610] | 0.152 [-0.327 to 0.631]
Statistical Analysis 1: Comparison: Academic Detailing (AD) Only vs AD + LEAP Combined; Test type: Superiority; Mean Difference (Net) = -0.0428, 95% CI 2-sided [-0.339 to 0.254]

ADVERSE EVENTS:
Time Frame: Adverse events were not monitored. Not applicable.
Description: Adverse events were not monitored. Not applicable.
Groups:
- Academic Detailing (AD) Only: Academic Detailing (AD): Site providers received one-on-one educational sessions between a non-physician professional trained in communication skills and the specific topic area (the Academic Detailer) aimed at increasing the use of the evidence-based practices. (PMID: 35568903)
- AD + LEAP Combined: Academic Detailing (AD): Site providers received one-on-one educational sessions between a non-physician professional trained in communication skills and the specific topic area (the Academic Detailer) aimed at increasing the use of the evidence-based practices. (PMID: 35568903) LEAP: Sites also received the Learn. Engage. Act. Process. (LEAP) program, which is a 6-month quality improvement coaching program plus a 6-month follow-up. (PMID: 32901440)
Arm/Group | Academic Detailing (AD) Only | AD + LEAP Combined
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This evaluation was developed by combining three smaller cluster randomized control trials on different topic areas. In the early post-coronavirus disease 2019 (COVID-19) era, site-level engagement was extremely difficult, perhaps minimizing the impact of the interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT05065502/Prot_SAP_000.pdf